CLINICAL TRIAL: NCT03037164
Title: Randomized, Double-Blind, Controlled, Parallel Group Study With the INTERCEPT Blood System for RBCs in Regions at Potential Risk for Zika Virus Transfusion-Transmitted Infections and Treatment Use Open-Label Extension Study
Brief Title: INTERCEPT Blood System for RBCs Study in Regions at Potential Risk for Zika Virus Transfusion-Transmitted Infections
Acronym: RedeS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI 00126
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Anemia
Keywords: INTERCEPT; Red Blood Cells; RBC; Pathogen Inactivation; Zika; Cerus; Pathogen Reduction
MeSH Terms: conditions — Anemia; Zika Virus Infection | interventions — Erythrocyte Count

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- INTERCEPT (Test) (Experimental): Red blood cell components treated with the INTERCEPT Blood System for Red Blood Cells ordered and administered to study patients by their treating physicians according to the local standards of care
  Interventions: Device: INTERCEPT Blood System for Red Blood Cells
- Conventional (Control) (Active Comparator): Conventional RBC components ordered and administered to study patients by their treating physicians according to the local standards of care
  Interventions: Device: Conventional (Control)

INTERVENTIONS:
Device: INTERCEPT Blood System for Red Blood Cells — The pathogen reduction process begins with a unit of RBCs derived from whole blood that is separated according to local regulations and standard operating procedures at the Blood Centers. RBCs are suspended in AS-5 or SAG-M for non-US sites. Leukocyte-reduction of whole blood or RBCs will be performed per manufacturer's instructions. The INTERCEPT Blood System process is performed on a single unit of leukocyte-depleted RBC in AS-5.
  Arms: INTERCEPT (Test)
Device: Conventional (Control) — Conventional RBC components ordered and administered to study patients by their treating physicians according to the local standards of care
  Arms: Conventional (Control)

SUMMARY:
Stage A: To evaluate the safety and efficacy of red blood cells (RBCs) prepared with the INTERCEPT Blood System for Red Blood Cells Pathogen Reduction Treatment (PRT) in comparison to conventional RBCs in patients who require RBC transfusion support.

Stage B: To provide early access to the INTERCEPT pathogen reduction system for RBC in regions where a substantial proportion of the population has been infected or is at risk of a transfusion-transmissible infection.

The objectives and design of Stage B will be reassessed on the completion of Stage A, in consultation with the FDA.

DETAILED DESCRIPTION:
Stage A

Patients will be approached, consented, screened for eligibility and randomized to receive either Test or Control RBCs in one of the three arms at the beginning of the study:

* Bleeding or non-bleeding patients at baseline may be enrolled into the 28-day transfusion period.
* Non-bleeding patients at baseline with chronic anemia requiring repeated simple transfusion may be enrolled into the 28-day +6-month extension period.
* SCD on a regular repeated RCE program at baseline may be enrolled into 28-day +6-month extension period to receive 3 consecutive RCE procedures.

Eligible patients will be randomized and transfused with study RBCs (Test or Control with 1:1 ratio) according to local practices for up to 28 days of transfusion support. Following the 28-day acute transfusion support period, patients will be transfused with conventional RBC components as indicated by their treating physician unless they were enrolled at baseline in the optional 6-month extension period.

Non-bleeding patients at baseline requiring repeated RBC transfusion for congenital or acquired chronic anemia (e.g., sickle anemia, thalassemia, other hemoglobinopathies, myelodysplastic syndrome, aplastic anemia, chemotherapy or stem cell transplant etc.) will be eligible to participate in an extension option for up to 6 months to evaluate patients requiring repeated transfusion for chronic anemia.

In addition, SCD patients on a regular RCE program at 2 or more clinical sites may be enrolled at baseline into the 6-month extension period to receive up to a total of 3 consecutive RCE procedures.

Screening/Recruitment

All potentially eligible patients at participating institutions will be approached for study consent. Subjects <18 years of age will require subject assent and parental consent. For subjects eligible for enrollment into the 6-month extension period option, consent/assent for the extension period should be obtained at initial enrollment.

Patients who consent to the study will be assigned a study ID number and undergo screening. Screening data collection and procedures will include:

Demographics (age, sex), vital signs, height, weight, indication for anticipated transfusion, type of scheduled surgery (if applicable), medical and surgical history, transfusion history, physical examination, comorbid conditions, concomitant medications, hematology panel (including complete blood count), blood type and Rh, Indirect Antiglobulin Test (IAT), blood chemistry, coagulation panel, Direct Antiglobulin Test (DAT), immune reactivity to IBS RBCs (if available), pregnancy test (when applicable). Once all screening assessments are completed and eligibility is confirmed, the subject may be randomized.

For SCD patients on a regular RCE program, if available in the medical record, the pre- and post- RCE total Hemoglobin, HbA, HbS and HgF concentrations should be recorded for up to 6 months prior to the first study transfusion.

If results from the following assessments are available in the medical record within 30 days prior to randomization, those data may serve as the screening data and the assessments do not need to be repeated unless the subject has an RBC transfusion in the 30-day period:

* hematology panel (complete blood count), blood chemistry and coagulation panel
* blood type and Rh
* IAT, DAT, and immune reactivity to IBS RBCs
* physical examination

If an RBC transfusion occurs after the study specific blood draws and assessments to determine eligibility are taken but prior to randomization, the subject may be randomized and the tests listed above should repeated prior to the first study transfusion.

A pregnancy test (when applicable) must be performed within 7 days of randomization.

Randomization and Blinding

For Stage A, potentially eligible patients will be consented and begin screening in the study in order to be assessed for eligibility for one of the three study arms and to be considered for randomization to receive Test or Control RBCs. An Interactive Web Response System (IWRS) will be used for electronic randomization of eligible patients.

Randomization will be at a 1:1 ratio of Test: Control to receive either Test or Control RBCs and stratified by site, baseline bleeding status [indication for RBC transfusion due to active bleeding (WHO Grade 3 or 4, APPENDIX 5) or for anemia without active bleeding], and participation of the optional extension period (yes/no). Anticipated surgical bleeding and planned blood loss/replacement through RCE at baseline should be included as active bleeding (Grade ≥3) by definition. Randomized patients who do not receive any study RBC transfusions through 28 days after randomization will be withdrawn from the study and replaced. Additional data will not be collected for these patients. These subjects may be reassessed for eligibility and re-enrollment after withdrawal.

At the end of screening, the patient's eligibility status will be entered into the electronic data capture system (EDC). If eligible, the patient will be randomized. Only appropriate blood bank staff will be able to access the treatment arm assignment. Study RBC unit labels will be indistinguishable for Test and Control products. Medical staff, and others caring for participating patients, as well as the sponsor (and delegates) will be blinded to treatment assignment. Unblinded delegates will monitor the production of the RBC components at designated blood centers.

Treatment

Randomized patients will be transfused with Test or Control RBC components for up to 28 days in the initial acute transfusion period and for an additional 6-months if the subject is entered into the optional extension period. Subjects participating in Stage A's optional extended study will continue to receive the same study article (Test or Control RBC) as in their initial 28-day study period. Following participation in the optional 6-month extended transfusion support period, patients will be transfused with conventional RBC components as indicated by their treating physician.

An RBC transfusion episode is defined to include consecutive RBC units transfused until the next post-transfusion Hb determination with ≤12 hours between transfusions (from the end of a prior component transfused to the start of a subsequent component transfused).

A confirmed negative immune reaction to IBS RBC is required prior to the first study transfusion and at every time point a Type/Rh and Screen (IAT) is performed for a patient within the 28-day acute transfusion period or during the extension period. Compatibility for RBC antigens will be confirmed using site's SOPs prior to transfusion of study RBCs. In case of confirmed physiologically active antibodies to IBS RBC or any presumed or documented antibodies to IBS RBC that preclude further transfusion with study RBCs, patients will be withdrawn from the study treatment and supported with conventional RBC components and followed for safety. Patients with antibodies to IBS RBC will be investigated for evidence of hemolysis and continue with all planned visits and safety monitoring.

SCD patients on a regular RCE program enrolled into the 6-month extension period will receive 3 consecutive RCE procedures with study RBC with an interval of 3-8 weeks between RCE procedures, as determined by their physician.

Study Assessments: Monitoring and Follow-up

Acute Transfusion Support Period (First study transfusion through Day 28 or death) and the optional extension period (if applicable).

The acute transfusion support period will comprise 28 days from the day of the first study transfusion (Day 1) through Day 28, or death of a patient, plus an additional optional 6-month transfusion period for those patients entered into the extension period. During these periods, patients will receive as many study RBCs as deemed appropriate by the treating physician. All AEs, SAEs, TRs and unanticipated adverse device effects will be collected starting from the initiation of the first study transfusion through 28 days after the last study transfusion. The Investigators will assess each AE/SAE/TR and unanticipated adverse device effects for relation to the transfused study RBCs. Transfusion reactions will be classified by the definitions in the CDC NHSN Hemovigilance Module Surveillance Protocol (APPENDIX 1, 2 & 3) and will be captured in the eCRF and, if in routine use, in the CDC NHSN Biovigilance Component/Hemovigilance Module (www.cdc.gov/nhsn).

Most proximate vital signs in the medical record will be collected prior to and following each study transfusion. The subject's hemoglobin value will be collected from the medical record, or if not available, a study sample will be submitted for testing, prior to and following each study transfusion episode within 15 minutes to 24 hours after the end of the transfusion episode and before the next RBC transfusion.

Relevant concomitant medications taken during the study and blood products transfused will be recorded with indication, total daily dose, and dates of drug administration.

During the acute transfusion support period, patients will undergo the following assessments prior to each transfusion episode: vital signs, AEs, TRs, SAEs and unanticipated adverse device effects, comorbid conditions, blood samples for safety labs (complete blood count, blood chemistry panel), IAT and immune reactivity to IBS RBCs. Samples may be used for additional in vitro research tests as required to confirm transfusion-transmitted pathogen mediated infections.

An immune reactivity to IBS RBCs test will be performed and resulted each time an IAT is performed within the 28-day acute and 6-month extension transfusion support period.

For SCD patients undergoing regular RCE, the following parameters should be assessed before and 15 mins to 4 hours after each RCE procedure:

* Complete blood count including Hb and reticulocytes; and proportion (%) of HbS, HbA, and HbF.
* Coagulation panel (INR, PT, aPTT).
* Plasma frozen sample for determination of S-300 and GSH concentrations.

Day 14 ±7 days after each RCE procedure for SCD patients undergoing regular RCE:

• Complete blood count including Hb and reticulocytes; and proportion (%) of HbS, HbA, and HbF.

Follow-Up Period (28 and 75 days after last study transfusion) for all transfused patients:

For the purposes of the Day 28 (± 7 days) and Day 75 (± 15 days) follow-up visits, Day 1 of the follow-up period is the day after the last study transfusion, either in the initial 28-day acute transfusion period or, if the subject is entered, in the optional extension period.

Day 28 (± 7 days) After the Last Study Transfusion (or before first post-study RCE with conventional RBCs in patients on a regular RCE program):

Vital signs will be collected, and blood samples will be collected for:

1. Routine safety labs (complete blood count, blood chemistry panel, hematology panel, and coagulation panel)
2. DAT and IAT
3. Immune reactivity test for IBS RBC
4. For SCD patients undergoing regular RCE:

   * Complete blood count including Hb and reticulocytes; and proportion (%) of HbS, HbA, and HbF.
   * Plasma frozen sample for determination of S-300 and GSH concentrations.

All AEs, SAEs, TRs and unanticipated adverse device effects will be reviewed and recorded for the period from the first study transfusion through 28 days after the last study transfusion.

End of Study Visit (Day 75 ±15 days) for all transfused patients:

Day 75 (± 15 days) after the last study transfusion either in the initial 28-day acute transfusion period or after the extension period, a blood sample will be collected for a DAT and immune reactivity test for IBS RBC.

ELIGIBILITY:
Stage A: Inclusion Criteria:

* Age ≥ 4 years.
* Patients who require or are expected to require a transfusion of RBC component(s), including red cell exchange transfusion
* Signed and dated informed consent form.
* Female patients of child-bearing potential must:

  * Have negative serum or urine pregnancy tests prior to study treatment to rule out pregnancy, and
  * Agree to use to use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner for the duration of study participation and an additional 28 days.

For 28-day +6-month extension study in chronically transfused patients:

• A diagnosis of a bone marrow failure syndrome requiring repeated RBC transfusion for congenital or acquired chronic anemia (e.g., sickle cell anemia, thalassemia, other hemoglobinopathies, myelodysplastic syndrome, aplastic anemia, chemotherapy or stem cell transplant etc.)

For 28-day +6-month extension study in SCD patients requiring regular repeated RCE.

* Diagnosis of SCD, either HbSS, HbSC or HbSB0 thalassemia, confirmed by Hb electrophoresis, deoxyribonucleic acid (DNA) analysis or high-performance liquid chromatography (HPLC)
* Currently participating in an automated RCE transfusion program (for at least 3 months prior to enrollment) with 3-to-8 week intervals between RCE transfusion episodes

Stage A: Exclusion Criteria

* Confirmed positive baseline serum/plasma antibody specific to IBS RBC (S 303 treated RBC) as determined by INTERCEPT S 303 antibody screening panel prior to receiving the first study transfusion
* Pregnant or breast feeding.
* Presence of an RBC warm autoantibody with evidence of active hemolysis.
* Positive DAT as defined below:

  * A polyspecific-DAT reaction strength > 2+, or
  * A polyspecific-DAT (any strength) in conjunction with pan-reactivity with a commercial IAT antibody screening panel that precludes the identification of underlying alloantibodies or indicates the presence of autoantibody.
* Have had an RBC transfusion within 7 days prior to randomization.
* Have received investigational products, including investigational blood products, pharmacologic agents or imaging materials, within 28 days prior to randomization. Prior receipt of conventional blood products tested with an investigational NAT test is not considered ground for exclusion.
* Patients presenting with or expected to have massive hemorrhage (≥10 RBC units within 24 hours) or expected to require massive transfusion protocols. Planned red cell exchange does not apply.
* Patients who require neonatal transfusions and intrauterine transfusions.
* Pre-existing antibody to RBC antigens that may make the provision of compatible study RBC components difficult.
* History of transfusion reactions requiring washed RBCs, volume reduced RBC, or RBCs with additive solution removed.
* Patients with documented IgA deficiency or a history of severe allergic reactions to blood products.
* For SCD patients to be enrolled into the repeated RCE 28-day +6-month arm of the study:

  * A history of acute chest syndrome in the last 6 months, or hyperhemolysis syndrome at any time.
  * Clinical evidence of splenic hyperfunction or splenic enlargement: ≥18 cm in longitudinal diameter (diagnosed at the Investigator's discretion according to the data available, with ultrasound data being preferable).
  * Currently receiving chemotherapy for treatment of cancer. Hydroxyurea for SCD is acceptable if subject has been on stable therapy for 3 months and no changes to dosage are planned.
  * Subject is in active treatment with renal dialysis.
  * Any subject for whom a substantial change in the number of RBC components transfused is anticipated due to anticipated splenectomy, bone marrow transplant, surgery or other change in clinical status.
  * Subject with known G6PD deficiency or requiring treatment with medications that are known to adversely affect RBC viability or bone marrow function.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adjusted hemoglobin increment | 15 minutes - 24 hours post transfusion
  The difference between the pre-transfusion and post transfusion episode hemoglobin values divided by the total hemoglobin content transfused, averaged over one or more transfusion episodes in patients without active bleeding at baseline (active bleeding is defined as WHO Grade 3 or 4 bleeding)
Adverse Events | 28 days
  Proportion of patients with any treatment-emergent adverse events (AEs) possibly, probably, or definitely related to study RBC transfusion through 28 days after the last study transfusion.
Treatment emergent antibodies | 75 days
  The proportion of patients with treatment emergent antibodies with confirmed specificity to IBS RBCs

SECONDARY OUTCOMES:
Adjusted hemoglobin consumption | 211 Days
  Defined as total hemoglobin mass transfused in grams divided by body weight in kg at baseline and duration of the study transfusion period in days (g/kg/day), in patients without active bleeding at baseline.
HbA clearance | 211 days
  HbA clearance in patients with SCD undergoing regular repeated RCE
Adverse Events | 28 Days after last study transfusion
  Treatment-emergent AEs
Transfusion reactions related to study RBCs (test or control) | 28 Days after last study transfusion
  Defined by the CDC National Healthcare Safety Network [NHSN] Hemovigilance Module protocol
RBC allo-antigens | 28 days
  Treatment-emergent immunization to RBC allo-antigens
Mortality | 28 Days after last study transfusion
  All-cause mortality
Adverse Events of Special Interest (AESI) | 28 Days after last study RCE
  Proportion of subjects with adverse events of special interest (AESI) through 28 days after the last study transfusion.
S-300 and GSH plasma levels | 15 minutes to 4 hrs after RCE
  S-300 and Glutathione (GSH) plasma levels

CONTACTS AND LOCATIONS:
Locations (16):
- United States (12):
  - Phoenix Children's Hospital (PCH), Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Grady Health System, Atlanta, Georgia
  - CHOA (Children's Healthcare of Atlanta), Atlanta, Georgia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - C4TKs (Cure 4 The Kids), Las Vegas, Nevada
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Versiti, Wauwatosa, Wisconsin
- Puerto Rico (3):
  - Menonita General Hospital, Aibonito
  - HIMA San Pablo Hospital, Caguas
  - San Juan Bautista School of Medicine Clinical Research Unit, Caguas
- Ege University Hospital, Izmir, Turkey (Türkiye)